CLINICAL TRIAL: NCT01916928
Title: The Use of Cell Free Fetal DNA in the Maternal Blood in the Evaluation of Intrauterine Fetal Demise and Miscarriage
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Sequenom Laboratories (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2012-414
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Results first posted 2015-02-02 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-02

CONDITIONS: Circulating Cell Free Fetal DNA; Intrauterine Fetal Demise; Miscarriage
Keywords: Circulating cell free fetal DNA; Intrauterine fetal demise; Miscarriage
MeSH Terms: conditions — Stillbirth; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection will consist of two ten milliliters samples of whole blood in the cffDNA STRECK tube. Plasma will be retained for analysis of circulating cell free fetal DNA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-viable pregnancy: Women presenting with stillbirth, defined as fetal death occurring after 20 weeks gestation or with miscarriage, defined as fetal death prior to 20 weeks gestation.

SUMMARY:
Women presenting to Washington Hospital Center with fetal loss would be offered participation in the study. The objective is to determine if ccffDNA obtained from maternal blood is present in the setting of missed abortion or fetal demise.

The investigators primary hypothesis is that cell free fetal DNA will be present in maternal blood in the presence of a failed pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with Intrauterine fetal demised or missed abortion

Exclusion Criteria:

* Patients diagnosed with threatened abortion with cardiac activity present
* Patients with IUFD who have delivered the fetus (the induction process may already be in process, however, the fetus and placenta must be in situ at the time of blood sampling)
* Patients with known genetic abnormalities or mental retardation as a result of chromosomal abnormalities 13, 18, 21, or sex chromosomes.
* Children under the age of 18
* Patients not fluent in or unable to consent to the study in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women presenting to Washington Hospital Center with fetal loss would be offered DNA sequencing of cell free fetal DNA from maternal blood in addition to the standard workup for fetal demise and miscarriage as deemed appropriate by the patient's care provider. Only women with sonographic evidence of products of conception in-utero will be offered enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita W Driggers, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Medstar Washington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Nagaishi M, Yamamoto T, Iinuma K, Shimomura K, Berend SA, Knops J. Chromosome abnormalities identified in 347 spontaneous abortions collected in Japan. J Obstet Gynaecol Res. 2004 Jun;30(3):237-41. doi: 10.1111/j.1447-0756.2004.00191.x. PMID 15210050
- [Background] Baena N, Guitart M, Ferreres JC, Gabau E, Corona M, Mellado F, Egozcue J, Caballin MR. Fetal and placenta chromosome constitution in 237 pregnancy losses. Ann Genet. 2001 Apr-Jun;44(2):83-8. doi: 10.1016/s0003-3995(01)01042-5. PMID 11522246
- [Background] Reddy UM, Page GP, Saade GR. The role of DNA microarrays in the evaluation of fetal death. Prenat Diagn. 2012 Apr;32(4):371-5. doi: 10.1002/pd.3825. PMID 22467168
- [Background] American Congress of Obstetricians and Gynecologists, Management of Stillbirth. ACOG Practice Bulletin, 2009. 102
- [Background] Palomaki GE, Kloza EM, Lambert-Messerlian GM, Haddow JE, Neveux LM, Ehrich M, van den Boom D, Bombard AT, Deciu C, Grody WW, Nelson SF, Canick JA. DNA sequencing of maternal plasma to detect Down syndrome: an international clinical validation study. Genet Med. 2011 Nov;13(11):913-20. doi: 10.1097/GIM.0b013e3182368a0e. PMID 22005709
- [Background] Kyle PM, Sepulveda W, Blunt S, Davies G, Cox PM, Fisk NM. High failure rate of postmortem karyotyping after termination for fetal abnormality. Obstet Gynecol. 1996 Nov;88(5):859-62. doi: 10.1016/0029-7844(96)00311-0. PMID 8885928
- [Background] MacDorman MF, Kirmeyer S. Fetal and perinatal mortality, United States, 2005. Natl Vital Stat Rep. 2009 Jan 28;57(8):1-19. PMID 19294965
- [Derived] Clark-Ganheart CA, Fries MH, Leifheit KM, Jensen TJ, Moreno-Ruiz NL, Ye PP, Jennings JM, Driggers RW. Use of cell-free DNA in the investigation of intrauterine fetal demise and miscarriage. Obstet Gynecol. 2015 Jun;125(6):1321-1329. doi: 10.1097/AOG.0000000000000863. PMID 26000503

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-viable Pregnancy
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis of cell free fetal DNA in 50 non-viable pregnancies.
Arm/Group | Non-viable Pregnancy
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age of participants.
  years | 31.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: The Presence or Absence of Cell Free Fetal DNA in Maternal Blood in the Setting of a Failed Pregnancy.
Description: Percentage of participants with the presence of cell free fetal DNA in maternal circulation after miscarriage of intrauterine fetal demise
Time Frame: During initial presentation for treatment
Measure: Number; unit: percentage of participants
Arm/Group | Non-viable Pregnancy
Number analyzed (Participants) | 50
percentage of participants | 50

2. Secondary Outcome: The Accuracy of ccffDNA Compared to Genetic Information Obtained From Amniocentesis, Chorionic Villus Sampling, Fetal, or Placental Tissue.
Time Frame: 3-4 weeks after specimen processing
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed as part of this study
Arm/Group | Non-viable Pregnancy
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No